CLINICAL TRIAL: NCT05024019
Title: A Multicenter Clinical Study of Nimotuzumab Combined With Concurrent Radiotherapy Versus Radiotherapy Alone in High-risk Patients With Head and Neck Squamous Cell Carcinoma Not Suitable for Cisplatin After Surgery
Brief Title: Nimotuzumab Combined With Radiotherapy in High-risk Patients With HNSCC Not Suitable for Cisplatin After Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPL-Nim-SCCHN-6
Record Dates: First submitted 2021-08-15; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Nimotuzumab; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group received nimotuzumab (200mg, weekly, for 6 weeks) combined with concurrent radiotherapy.
  Interventions: Drug: Nimotuzumab
- Control group (No Intervention): The control group received radiotherapy alone.

INTERVENTIONS:
Drug: Nimotuzumab — The study group received nimotuzumab (200mg, weekly, for 6 weeks) in combination with radiotherapy.
  Arms: Study group

SUMMARY:
This study is a prospective, open label, multicenter, randomized controlled clinical trial. The main purpose of the study is to evaluate the efficacy and safety of nimotuzumab combined with concurrent radiotherapy versus radiotherapy alone in high-risk patients with HNSCC not suitable for cisplatin after surgery. The subjects were randomly divided into study group (nimotuzumab combined with concurrent radiotherapy) and control group (radiotherapy alone) by 1∶1 stratified random method.

DETAILED DESCRIPTION:
This study is a prospective, open label, multicenter, randomized controlled clinical trial. The main purpose of the study is to evaluate the efficacy and safety of nimotuzumab combined with concurrent radiotherapy versus radiotherapy alone in high-risk patients with HNSCC not suitable for cisplatin after surgery. The subjects were randomly divided into study group and control group by 1∶1 stratified random method. The study group received nimotuzumab (200mg, weekly, for 6 weeks) combined with concurrent radiotherapy, while the control group received radiotherapy alone. The main endpoint is 2 year disease free survival (DFS) rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histology or imaging diagnosed as head and neck (oropharyngeal cancer, hypopharyngeal cancer, laryngeal cancer) squamous cell carcinoma; oropharyngeal cancer should be p16 negative (p16 positive defined as p16 ≥ 70%);
3. The radical surgery has been completed and patients were suffered from any postoperative risk factors as follows: (1) extranodal extension (ENE); (2) pT3-4; pN2-3; (3) Nerve invasion (PNI) or vascular invasion (LVI); (4) Lymph node metastasis in zone IV or zone V (oral/oropharyngeal cancer); (5) Proximal margin (< 5mm);
4. Immunohistochemical detection indicated the EGFR expressions were positive;
5. The patients were not suitable for cisplatin chemotherapy: (1) Age>65 years; (2) ECOG PS score>2; (3) Renal dysfunction (creatinine clearance <60ml/min); (4) Severe tinnitus or hearing loss (need hearing aids or hearing tests show 25 decibels threshold or above at two consecutive frequencies); (5) peripheral neuropathy severer than 1 level ; (6) Unable to accept venous hydration, such as cardiac dysfunction or other comorbidities (judged by the investigator); (7) The patient refuses cisplatin chemotherapy;
6. Imaging examination did not suggest distant metastasis;
7. Expected survival time ≥ 6 months;
8. The following criteria must be met (No transfusion of blood or blood products within 14 days prior to screening): Hb≥90g /L; ANC≥1.0×10*9 /L; PLT≥80×10*9 /L; white blood cell count ≥ 4×10*9 /L; Biochemical examination need to meet the following criteria: serum total bilirubin (TBIL) ≤1.5 ULN; aminotransferase (AST)/alanine aminotransferase (ALT) ≤2.5 ULN.
9. For females of reproductive age, the patients must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment and be willing to use a reliable method of contraception during the trial. Male subjects should use a reliable method of contraception from the beginning of treatment until 120 days after the last medication;
10. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up.

Exclusion Criteria:

1. The patients received chemotherapies, PD-1 inhibitors, monoclonal antibody against EGFR, EGFR-TKI, anti-angiogenic drugs within 4 weeks before enrollment;
2. The patients participated in other interventional clinical trials within 30 days before screening;
3. There was a history of other malignant tumors within the past 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ;
4. Poorly controlled concurrent diseases (such as heart failure, diabetes, hypertension, thyroid disease, mental illness, etc.);
5. Known to be infected with HIV virus or active viral hepatitis or tuberculosis;
6. There is major surgery within 30 days before taking the trial drug for the first time or there is planned surgery;
7. Allergic to the drugs or their components used in this program;
8. Pregnancy (confirmed by blood or urine HCG test) or breastfeeding women, or subjects of childbearing age who are unwilling or unable to take effective contraceptive measures (applicable to both male and female subjects) until at least 6 months after the last trial treatment;
9. Patients who are not suitable to participate in this research according to the evaluations of researchers;
10. Those who are unwilling to participate in this study or unable to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2021-08-21 (Estimated); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-08-21 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 2 year

SECONDARY OUTCOMES:
Overall survival (OS) | 2 year
Local area recurrence free survival (LRRFS) | 2 year
Distant metastasis free survival (DMFS) | 2 year
Quality of life assessed by EORTC QLQ-H&N35 | 2 year
  Quality of life assessed by EORTC QLQ-H&N35 [EORTC QLQ-H&N35 is a specific quality of life assessment scale based on EORTC QLQ-C 30, with 35 items. All of the scales and single-item measures range from 0 to 100. A high score represents a higher response level.]
Incidence of treatment-emergent adverse events | 2 year
  Including the incidence of treatment-emergent adverse events[Safety and Tolerability]. Adverse events should be reported and graded according to CTCAE version 5.0.

OTHER OUTCOMES:
The change of tumor related markers | 2 year
  The correlation of the value of EGFR, SCC-Ag, CEA and therapeutic effect [The changes of serum tumor markers (such as SCC-Ag and CEA were observed before and after treatment. The baseline EGFR levels on the prognosis of patients should also be explored]

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Jiangsu Province Hospital, Nanjing
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shanghai General Hospital/First People's Hospital Affiliated with Shanghai Jiao Tong University, Shanghai